CLINICAL TRIAL: NCT04909203
Title: iKinnect2.0 for Juvenile Justice Involved Youth at Risk for Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R44MH126819 (NIH); R44MH126819 (NIH)
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Child Behavior Disorders; Suicide and Self-harm
Keywords: Criminal Justice; Juvenile Delinquency; Adolescent Suicidality; Self-Help Device; Assistive Technology
MeSH Terms: conditions — Child Behavior Disorders; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iKinnect2.0 (Experimental): Parent-Youth dyads assigned to the iKinnect2.0 condition will be given access to the iKinnect2.0 app that has been developed for this study. Parent and youth will be asked to download the app to their phone during the baseline assessment process and asked to use it as often as they would like throughout the duration of the 16 week trial. The app is designed to be used several times throughout each day.
  Interventions: Device: iKinnect2.0
- Attention-Control Placebo App & Supporting Materials (Placebo Comparator): Parent-Youth dyads assigned to the control condition will be asked to download the free Life360 app to their phone during the baseline assessment process and will also be given access to an online suicide resources brochure. Participants will be asked to use the control-condition app and associated materials as often as they would like throughout the duration of the 16 week trial.
  Interventions: Device: Active Control App

INTERVENTIONS:
Device: iKinnect2.0 — iKinnect2.0 is a paired mobile phone app for use on both Android and iOS operating systems by youth with conduct disorders and their parents.
  Arms: iKinnect2.0
Device: Active Control App — Mobile phone app for use on both Android and iOS operating systems for GPS tracking of other persons.
  Arms: Attention-Control Placebo App & Supporting Materials

SUMMARY:
This study is a 16-week intent-to-treat randomized controlled trial (RCT) with 120 suicidal juvenile justice (JJ)-involved transition-age (TA) youth (age 15-21 years) and a primary caregiver (dyads). Dyads will be randomly assigned to iKinnect2.0 (n=60 dyads) or Life360 (control app) plus an electronic suicide resources brochure (n=60 dyads). This design will test iKinnect2.0's new features for suicide prevention against TA youth awareness of and access to high-quality suicide prevention resources, while simultaneously testing features relating to conduct problems and parent management against parents knowing the TA youth's whereabouts in real-time and controlling for dyad member engagement in technology (Life360). Participants will be assessed at baseline, 4, 8 and 16 weeks. Primary youth-reported outcomes relating to suicide risk include: Suicidal behaviors (ideation, planning, attempts), non-suicidal self-injurious behaviors, self-efficacy in coping with distress, and use of imminent distress coping strategies (behavioral skills, use of crisis stabilization plan). Youth will also report on their criminal behavior. Primary caregiver-reported outcome variables relating to youth suicide include: Self-efficacy in applying family-based suicide-prevention strategies and reported use of those strategies; caregivers will also report on their own functioning (efficacy/confidence in parenting skills, life stress), TA youth functioning (internalizing and externalizing symptoms), parental management behaviors (expectation clarity, parental monitoring, discipline effectiveness/consistency, use of rewards), and parent-youth relationship quality (communication, conflict, support). App satisfaction and use of technology outcomes (i.e., degree of app usage, features used) will be examined and reported descriptively.

DETAILED DESCRIPTION:
The goal of this 33-month Fast Track study is to significantly expand iKinnect, an efficacious paired mobile app that supports parents (in delivering) and youth (in receiving) evidence-based techniques to reduce youth problem behaviors such as delinquency and drug use. iKinnect2.0 will be expanded to also prevent non-suicidal self-injury (NSSI), suicidal behaviors, and death by suicide in juvenile justice (JJ) involved youth while continuing to prevent criminal recidivism. iKinnect was originally designed based on Multisystemic Therapy (MST) principles to help youth with serious conduct problems. Results from a randomized controlled trial (RCT; N=72) demonstrated its efficacy in reducing externalizing behaviors and improving parent effectiveness. This project seeks to significantly expand iKinnect to prevent NSSI, suicidal behaviors (ideation, planning, attempts), and death by suicide in JJ-involved transition age (TA) youth while continuing to decrease externalizing behaviors and prevent recidivism. Usability and acceptability testing will be conducted to test new features with target end-users (youth and their parents/guardians) and key stakeholders (probation officers, parole/re-entry officers, administrators, people with lived experience). Once usability and acceptability is achieved, an eight-week pilot will be conducted to test study procedures followed by a 16-week randomized controlled trial comparing iKinnect2.0 to an active control mobile app. Investigators expect that iKinnect2.0 participants will report a significantly greater decrease in youths' suicidal, NSSI, and conduct-problem behaviors, and less recidivism. Furthermore, iKinnect2.0 participants will report significantly greater use of behavioral skills and suicide prevention strategies (TA youth and parents), and greater self-efficacy in coping with emotional distress (TA youth). iKinnect2.0 parents will report greater awareness of and confidence in applying evidence-based strategies to prevent suicide/NSSI and to support their TA youth through a suicide crisis.

Investigators hypothesize that in comparison to the active control condition, iKinnect participants will show significantly better outcomes from baseline to the 4, 8, and 16-week assessment points such that:

1. iKinnect parents will report greater increases in parenting and suicide prevention efficacy.
2. iKinnect youth will report greater decreases in suicidal, NSSI, and delinquent/criminal behaviors.
3. iKinnect youth will report greater increases in coping with imminent distress and use of suicide prevention coping strategies.
4. iKinnect parents and youth will report greater increases in clarity of expectations, parental monitoring, discipline effectiveness, parent consistency, use of rewards, and positive parent-youth relations.
5. iKinnect parents will report greater decreases in youth problem behaviors.

ELIGIBILITY:
PARENT/GUARDIAN INCLUSION CRITERIA:

* 18 years or older
* Fluent in English
* Owns an Android or iPhone-based smartphone with a data plan and is the primary user of the phone
* Primary caregiver and supervisor of a youth aged 15-21 on probation or receiving post-incarceration reentry services at time of screening

YOUTH INCLUSION CRITERIA:

* Age 15-21 years
* Fluent in English
* Possesses and is the primary user of an Android or iPhone-based smartphone with a data plan
* Currently resides in same household as linked parent/legal guardian at least 5 days per week
* Has been arrested at least once and is receiving community-based JJ services related to probation or re-entry
* At significant risk for suicide, as evidenced by one of the following: one or more lifetime suicide attempts; elevated past-month suicidal ideation (>24 on the SIQ-JR99, or self-injury repetition (>3 lifetime self-harm episodes, including one in the past 12 weeks before screening)
* Willing to disclose NSSI and suicidal behaviors to parent

To ensure consistency of planned and actual enrollment, particularly of Black youth, researchers will begin to exclude youth of certain races once pre-established recruitment milestones for a specific racial group is achieved.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Suicidal Ideation Questionnaire Junior (SIQ-JR) | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses youth frequency of suicidal ideation Scores range from 0 to 90, with a published clinical cut-off score of 31. Higher aggregated scores indicate negative outcomes.
Change in Service Assessment for Children and Adolescents | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Interviewer-based structured measure to assess health care utilization with parallel parent and child versions. Parents report their children's mental health service-use history. Asks a maximum of 331 questions on service use by child (plus 10 introductory demographic questions). The initial 24 of the 331 are 'gate-level' questions which ask the parent about the child's lifetime use covering 23 different categories of service. A positive response on any lifetime service-use for a particular category leads to a separate section that askes more in-depth questions about service use in the past 12 months.
Change in Suicide Attempt Self-Injury Interview | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Interviewer-administered instrument to assess the occurrence of youth suicidal and non-suicidal self-injuries (frequency, intent, medical severity, and outcomes). The final measure is assessed for reliability and validity with collateral measures. This interview based
Change in Center for Epidemiological Studies-Depression Scale (CES-D) | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses self-reported depressive symptoms experienced. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
Change in The Coping Skills Use | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses frequency of skills use, perceived helpfulness of skills, and self-efficacy in using them. With 17 questions and responses ranging from 0 (strongly agree) to 4 (strongly disagree) there is a possible range of 0-68, with lower scores indicating better coping.
Change in Self-Report of Delinquency and Crime | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses frequency of youth engagement in particular delinquent or criminal behaviors. The 26-item widely-used measure asks youth to report how many times in the past two weeks they engaged in a number of delinquent and illegal behaviors. Total numbers of times are tallied for all items for the general delinquency scale (higher score indicates more delinquency). In addition, two subscales, status offenses and school delinquency may be examined.
Change in Achenbach (Child/Adult) Behavior Checklist | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses youth behavioral and emotional problems. Administered to parent only. Each subscale item relating to aggressive behavior (19 items; e.g., "gets in fights;" "attacks people") and rule breaking (17 items; e.g., "sets fires;" "steals outside of the home") had three possible responses (0=Not True; 1=Somewhat or sometimes true; 2=Very true or often true). With 113 questions and 3 spots for not covered behaviors a total possible range of 0 to 232; higher numbers indicate more problematic behaviors.
Change in Loeber Parenting Scale | baseline (time1), 1-4 weeks (time 2), 5-8 weeks (time 3), and 9-16 weeks (time 4)
  Assesses parent and youth clarity of expectations, discipline consistency/effectiveness, and use of rewards. With 25 questions and each subscale having 3 possible responses - Never, Sometimes, and Always. Possible range of scores for the whole set includes high prevalence or infrequency of negative parenting skills in supervision, discipline consistency, discipline effectiveness, and positive parenting subscales; higher scores equal higher prevalence, lower scores equal infrequency.
Change in app Satisfaction Survey | 1-16 weeks (time 4)
  Assess ease of use and helpfulness of the assigned app. With a parent and child version and 10 questions with answers ranging from 0 (strongly disagree) to 5 (strongly agree) there is a possible range of 0-50 for the question set with higher numbers indicating better user experience/outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Dimeff, PhD, Principal Investigator — Evidence-Based Practice Institute; Cindy Schaeffer, PhD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Evidence-Based Practice Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Requests for use of data will be considered on a case-by-case basis. Interested researchers may send data requests to research@ebpi.org